CLINICAL TRIAL: NCT04524169
Title: Immunotherapy for Elderly Patients With Chronic Osteoporotic Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OP pain - Immunotherapy
Record Dates: First submitted 2020-08-11; First posted 2020-08-24 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Osteoporotic Pain
Keywords: osteoporotic pain; Thymosin alpha 1
MeSH Terms: interventions — Thymalfasin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thymosin Alpha 1 (Experimental): Thymosin Alpha 1 will be subcutaneous injected to the participants twice per week for 4 weeks.
  Interventions: Drug: Thymosin Alpha1
- Standard Care (No Intervention): Participants under the regularly treatment

INTERVENTIONS:
Drug: Thymosin Alpha1 — Thymosin Alpha 1 will be subcutaneous injected to the participants twice per week for 4 weeks.
  Arms: Thymosin Alpha 1

SUMMARY:
Osteoporotic pain is the most common clinical symptom in elderly patients. The course of pain is prolonged and the effect of clinical treatment is limited. This study will observe the therapeutic effect of thymosin alpha 1 on elderly patient with osteoporotic pain and explore its immunotherapy mechanism.

DETAILED DESCRIPTION:
About 70% of the elderly patients suffered osteoporotic pain, mainly involving the limbs and low back. The pain prolonged and varies from mild to severe, and the effect of the clinical treatment is poor which has become a serious social problem. Recent studies have put forward a new point of "bone Immunology", which suggests that immune system, especially CD4+ T cell system, are involved in the regulation of bone formation, bone resorption and bone remodeling. So, in this study, the investigators will observe the therapeutic effect of thymosin alpha 1 on osteoporotic pain in elderly by observing the improvement of VAS score before and after the treatment, as well as the changes of proportion of peripheral blood CD4+ T lymphocyte subsets, bone mineral density, serum bone biochemical index, neuropeptides, RANKL and other cytokines levels will be evaluated. The clinical safety of thymosin alpha 1 in elderly patients with osteoporotic pain will also be observed.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffered osteoporotic pain diagnosed by specialists
* VAS scores greater than 5
* Normal reading and understanding ability
* Communicate normally
* Volunteer to participate

Exclusion Criteria:

* Mental illness
* Serious physical disease
* Unwilling to cooperate

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of VAS scores | 4 week
  The VAS (visual analogue scale) is a scale used to determine the pain intensity experienced by individuals. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain", "0" means no pain, "10" means severe worst pain. In our study VAS score will be record before and after 4 weeks of treatment.

SECONDARY OUTCOMES:
Change of BMD value | 4 week
  A bone mineral density (BMD) test is an easy, reliable test that measures the thickness of the bones and the response to osteoporosis treatment. We perform the BMD test by X-rays and record participants' BMD values before and after 4 weeks of treatment.

OTHER OUTCOMES:
Change of The CD4+ T-lymphocyte profile in peripheral blood | 4 week
  Lymphocytes in peripheral blood were isolated from participants before and after 4 weeks of treatment. The CD4+ T-lymphocyte profile was analyzed by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Yu, Study Chair — Department of Anesthesiology, Renji Hospital, School of Medicine, SJTU
Locations (1):
- Diansan Su, Shanghai, Shanghai Municipality, China